CLINICAL TRIAL: NCT06895460
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial on the Treatment of Bronchial Asthma With Budesonide Formoterol Combined With Immune Modulators (Staphylococcus and Neisseria Tablets)
Brief Title: A Trial on the Treatment of Bronchial Asthma With Budesonide Formoterol Combined With Immune Modulators (Staphylococcus and Neisseria Tablets)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL-BA-QIP-1001
Record Dates: First submitted 2025-02-27; First posted 2025-03-26 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Adjuvants, Immunologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide Formoterol combined with placebo (Placebo Comparator)
  Interventions: Drug: Budesonide Formoterol; Drug: Placebo
- Budesonide Formoterol Combined with Immune Modulators (Staphylococcus and Neisseria Tablets) (Experimental)
  Interventions: Drug: Budesonide Formoterol; Drug: Immune Modulators (Staphylococcus and Neisseria Tablets)

INTERVENTIONS:
Drug: Budesonide Formoterol — Investigator Selection
Drug: Placebo — Placebo: 0.3 mg/tablet, 4 tablets per dose, 3 times per day, for a course of 3 months
  Arms: Budesonide Formoterol combined with placebo
Drug: Immune Modulators (Staphylococcus and Neisseria Tablets) — Staphylococcus and Neisseria Tablets: 0.3 mg/tablet, 4 tablets per dose, 3 times per day, for a course of 3 months
  Arms: Budesonide Formoterol Combined with Immune Modulators (Staphylococcus and Neisseria Tablets)

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial on the Treatment of Bronchial Asthma with Budesonide Formoterol Combined with Immune Modulators (Staphylococcus and Neisseria Tablets)

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter clinical trial. A total of 198 participants with bronchial asthma are planned to be enrolled and randomized in a 1:1 ratio to the experimental group and the control group. The experimental group will receive Budesonide Formoterol Powder for Inhalation plus immune modulators (Staphylococcus and Neisseria Tablets), while the control group will receive Budesonide Formoterol Powder for Inhalation plus placebo. The treatment period is 3 months for both groups, followed by a 3-month follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 years, male or female;
2. Confirmed diagnosis of asthma at least 6 months prior to screening;
3. Patients with uncontrolled asthma (according to the 2024 GINA guidelines-asthma control level classification criteria, patients with partially controlled and uncontrolled asthma);
4. Within the past 6 months, at least one of the following positive test results for lung function:

   * Positive bronchodilator test with an increase in FEV1 of ≥12%, and an absolute increase in FEV1 of ≥200 ml;
   * Positive bronchial provocation test or exercise challenge test;
   * Peak expiratory flow (PEF) variability over 2 weeks with a daily variation rate of ≥20% or a weekly average variation rate of ≥10%;
   * Significant improvement in lung function after 4 weeks of asthma treatment, with an increase in FEV1 of ≥12%, an absolute increase in FEV1 of ≥200 ml, or an improvement in PEF of ≥20%;
5. Before the first administration of the study drug, the patient has good function of major organs and no contraindications to ICS + LABA treatment;
6. The participant (or their legal representative) must sign and date the informed consent form, indicating their understanding of the study's purpose and the procedures involved, and their willingness to participate in the study.

Exclusion Criteria:

1. Patients with a history of severe asthma (according to the definition in the Guidelines for the Prevention and Treatment of Bronchial Asthma (2024 Edition));
2. Patients in the acute exacerbation phase who may require intravenous/oral corticosteroids;
3. Patients with rheumatology and immunology conditions;
4. Atypical asthma or comorbidities such as pulmonary tuberculosis, chronic obstructive pulmonary disease, bronchiectasis, pulmonary embolism, severe respiratory failure, or other respiratory system diseases;
5. Individuals with significant diseases other than bronchial asthma. Significant diseases are defined as conditions that, in the investigator's judgment, may place the participant at risk or affect the study results, such as severe cardiovascular, cerebrovascular, hepatic, renal, hematologic diseases, malignancies, psychiatric disorders, immune system diseases, or pulmonary organic functional impairments;
6. Individuals allergic to the study drug or corticosteroids;
7. Participation in another clinical trial within 30 days prior to screening or currently ongoing;
8. Use of immune modulators (including thymosin, thymopeptides, interferon, transfer factor, Bacillus Calmette-Guérin polysaccharides, any type of bacterial extracts, such as Biostim, bacterial lysate capsules) within 30 days prior to the use of the study drug or during the study period;
9. Women who are currently pregnant or breastfeeding, or women of childbearing potential who cannot use contraception during the study period;
10. The participant is deemed unsuitable for study observation by the investigator.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The overall asthma control rate at 12 weeks of treatment | week 12
  The overall control rate = (number of well-controlled cases + number of partially controlled cases) / total number of cases × 100%

SECONDARY OUTCOMES:
The overall asthma control rate at 24 weeks of treatment | week 24
  The overall control rate = (number of well-controlled cases + number of partially controlled cases) / total number of cases × 100%
Number of acute asthma exacerbations | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Changes in Asthma Control Test (ACT) scores | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  The minimum and maximum scores of the Asthma Control Test are 5 and 25 points respectively. The higher the ACT score, the better the asthma control.
Changes in lung function indicators compared to baseline | Month 3, Month 6
  Changes in PEF
Five-point Asthma Quality of Life Scoring | Month 3, Month 6
  The minimum and maximum total scores of the 5-point asthma quality of life assessment are 35 and 175 points respectively. The higher the score, the better the patient's quality of life.
Adverse events (AEs) | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No